CLINICAL TRIAL: NCT04026399
Title: Neuroplasticity With Daily Use of a Sensorimotor Priming Vibration System to Improve Hand Function After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00086207; P20GM109040 (NIH)
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: Stroke; Physical Disability
Keywords: physical stimulation; Subliminal stimulation; stroke rehabilitation; upper extremity; paresis; hand function; occupational therapy; physical therapy
MeSH Terms: conditions — Stroke; Paresis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stimulation + therapy (Experimental): The participant receives stimulation and home therapy.
  Interventions: Other: peripheral vibration stimulation; Behavioral: therapy
- no stimulation + therapy (Sham Comparator): The participant receives no stimulation and receives home therapy.
  Interventions: Behavioral: therapy

INTERVENTIONS:
Other: peripheral vibration stimulation — wearing a wristband that delivers imperceptible vibratory stimulation.
  Arms: stimulation + therapy
Behavioral: therapy — practice of daily living tasks

SUMMARY:
More than 4 million stroke survivors in the U.S. suffer from post-stroke sensorimotor hand disability, which is typically permanent and difficult to treat. Hand disability has a profound negative impact on functional ability and independence. One way to improve hand function is to use peripheral sensory stimulation. Sensory stimulation in conjunction with therapy has been shown to improve motor outcomes more than therapy alone. While promising, most modalities of sensory stimulation interfere with natural hand tasks. To address these practical limitations, we have developed a new stimulation, imperceptible random-frequency vibration applied to wrist skin via a watch. In this study, we will determine if use of this vibration increases hand functional recovery.

DETAILED DESCRIPTION:
The study design is a double-blinded randomized controlled study. Subjects will wear the device for at least 8 hours/day every day for a month, during which they will come to the laboratory for weekly evaluation. Follow-up evaluation will occur 3 months after. The device will deliver vibration (treatment) or no vibration (control).

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke survivor (>= 6 months post stroke)
* Ability to move an object with the paretic hand
* Fingertip sensory deficits
* Ability to put on a watch daily (by oneself or with help)

Exclusion Criteria:

* Currently undergoing other upper extremity rehabilitation therapy
* Upper limb botulinum toxin within 3 months prior to or during enrollment
* Change in neurological disorder medications during the enrollment
* Complete upper limb deafferentation
* Rigidity (Modified Ashworth Scale=5)
* Brainstem stroke
* Comorbidity (peripheral neuropathy, orthopaedic conditions in the hand that limit ranges of motion, premorbid neurologic conditions, compromised skin integrity of the hand/wrist due to long-term use of blood thinners)
* Language barrier or cognitive impairment that precludes following instructions and/or providing consent

If a participant has contraindications for Transcranial Magnetic Stimulation (TMS), the participant will not do TMS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kautz, PhD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Caorlina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Scronce G, Ramakrishnan V, Vatinno AA, Seo NJ. Effect of Self-Directed Home Therapy Adherence Combined with TheraBracelet on Poststroke Hand Recovery: A Pilot Study. Stroke Res Treat. 2023 Mar 8;2023:3682898. doi: 10.1155/2023/3682898. eCollection 2023. PMID 36936523

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stimulation + Therapy | no Stimulation + Therapy
Started | 6 | 6
Completed | 1 | 3
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stimulation + Therapy | no Stimulation + Therapy | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12) | 61 (9) | 61 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Short-latency Afferent Inhibition
Description: motor evoked potential suppression by conditioning electrical stimulation
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: % of unconditioned motor evoked potentia
Arm/Group | Stimulation + Therapy | no Stimulation + Therapy
Number analyzed (Participants) | 3 | 2
% of unconditioned motor evoked potentia | 48 (56) | 21 (35)

2. Secondary Outcome: Action Research Arm Test
Description: standardized clinical upper extremity function score
Time Frame: 1 month
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Stroke Impact Scale Hand Subscale
Description: standardized patient-reported hand function assessment
Time Frame: 1 month
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Stoke Impact Scale Hand Subscale
Description: standardized patient-reported hand function assessment
Time Frame: 4 month
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Timing of Reactive Force Generation Per Perturbation
Description: time of reactive force
Time Frame: 1 month
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Timing of Reactive Force Generation Per Perturbation
Description: time of reactive force
Time Frame: 4 month
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Fugl-Meyer Upper Limb Assessment
Description: standardized clinical upper extremity function score
Time Frame: 1 month
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Fugl-Meyer Upper Limb Assessment
Description: standardized clinical upper extremity function score
Time Frame: 4 month
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Grip Force Direction
Description: angle of the grip force vector from the normal direction
Time Frame: 1 month
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Grip Force Direction
Description: angle of the grip force vector from the normal direction
Time Frame: 4 month
Reporting Status: Not Posted

11. Other Pre Specified Outcome: In-home Hand Use Amount
Description: affected hand use amount as measured by accelerometers
Time Frame: 1 month
Reporting Status: Not Posted

12. Other Pre Specified Outcome: In-home Hand Use Amount
Description: affected hand use amount as measured by accelerometers
Time Frame: 4 month
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Reactive Force Magnitude Per Perturbation
Description: magnitude of reactive grip force
Time Frame: 1 month
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Reactive Force Magnitude Per Perturbation
Description: magnitude of reactive grip force
Time Frame: 4 month
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Safety Margin
Description: additional force used during grip
Time Frame: 1 month
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Safety Margin
Description: additional force used during grip
Time Frame: 4 month
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Corticomotor Excitability
Description: motor evoked potential amplitude
Time Frame: 1 month
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Corticomotor Excitability
Description: motor evoked potential amplitude
Time Frame: 4 month
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Spectral Power Perturbation During Grip
Description: EEG spectral power perturbation during grip
Time Frame: 1 month
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Spectral Power Perturbation During Grip
Description: EEG spectral power perturbation during grip
Time Frame: 4 month
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Connectivity
Description: EEG coherence within the sensorimotor network
Time Frame: 1 month
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Connectivity
Description: EEG coherence within the sensorimotor network
Time Frame: 4 month
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Short-latency Afferent Inhibition
Description: motor evoked potential suppression by conditioning electrical stimulation
Time Frame: 4 month
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Box and Block Test
Description: number of blocks moved in a minute
Time Frame: 1 month
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Box and Block Test
Description: number of blocks moved in a minute
Time Frame: 4 month
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Wolf Motor Function Test
Description: standardized clinical upper extremity function score
Time Frame: 1 month
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Wolf Motor Function Test
Description: standardized clinical upper extremity function score
Time Frame: 4 month
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Action Research Arm Test
Description: standardized clinical upper extremity function score
Time Frame: 4 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Stimulation + Therapy | no Stimulation + Therapy
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stimulation + Therapy (N=6) | no Stimulation + Therapy (N=6)
gallbladder removal (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stimulation + Therapy (N=6) | no Stimulation + Therapy (N=6)
increased muscle tone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04026399/Prot_SAP_001.pdf
  • Informed Consent Form (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT04026399/ICF_000.pdf